CLINICAL TRIAL: NCT04187157
Title: Association Between the Implantation of Conventional or Blue Light-filtering Intraocular Lens and Survival Among Patients Undergoing Bilateral Cataract Surgery: a Multi-center, Observational Cohort Study
Brief Title: Association Between Light Spectrum and Survival After Cataract Surgery
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Matthew Rosengart, Professor, University of Pittsburgh
Other Study IDs: PRO18060034
Record Dates: First submitted 2019-11-26; First posted 2019-12-05 (Actual); Last update posted 2019-12-05 (Actual); Status verified 2019-12

CONDITIONS: Cataract; Age-related Cataract; Circadian Rhythm Disorders; Glaucoma; Age Related Macular Degeneration
Keywords: circadian; cataracts; blue light; survival
MeSH Terms: conditions — Cataract; Chronobiology Disorders; Glaucoma; Macular Degeneration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (2):
- Blue-light filtering intraocular lens (IOL): Bilateral implantation of blue-filtering intraocular lens. Blue-IOL, in addition to ultraviolet, also impede the transmission of the lower visible blue spectrum between 400 and 500nm.
  Interventions: Device: Blue-light filtering intraocular lens
- Conventional intraocular lens (IOL): Bilateral implantation of conventional ultraviolet light-blocking intraocular lens
  Interventions: Device: Conventional intraocular lens

INTERVENTIONS:
Device: Blue-light filtering intraocular lens — Bilateral implantation of blue light-blocking intraocular lens
  Groups: Blue-light filtering intraocular lens (IOL)
Device: Conventional intraocular lens — Bilateral implantation of conventional intraocular lens
  Groups: Conventional intraocular lens (IOL)

SUMMARY:
This study was a retrospective observational cohort analysis of subjects aged 65 years and older, who underwent bilateral cataract surgery within a single (15 hospital) healthcare system, to determine the association between type (conventional or blue-light filtering) of implanted intraocular lens and survival.

ELIGIBILITY:
Inclusion Criteria:

* The study population consisted of all adult patients (at least 65 years) who underwent bilateral cataract surgery between January 01, 2012 and January 01, 2018 within the University of Pittsburgh Medical Center (UPMC) healthcare system. To be considered bilateral and concomitant, cataract surgery had to be performed on both the left and the right eye within a 365-day period.

Exclusion Criteria:

* We excluded patients undergoing unilateral cataract surgery, surgery to replace or repair a previously implanted IOL, or bilateral implantation with one Blue-IOL and one Natural-IOL (i.e., mixed IOL transmission properties).

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: The study population consisted of all adult patients (at least 65 years) who underwent bilateral cataract surgery between January 01, 2012 and January 01, 2018 within the University of Pittsburgh Medical Center (UPMC) healthcare system.
Sampling Method: Non-Probability Sample
Enrollment: 10192 (Actual)
Dates: Start 2012-01-01 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-04-30 (Actual)

PRIMARY OUTCOMES:
All-cause mortality | From the date of the initial cataract surgery until the date of death or end of the study period (April 30, 2019), whichever occurred first, assessed up to 2,310 days.
  The primary outcome was all-cause mortality. Mortality was identified based on the Social Security Death Master File and discharge status. Follow-up started from the day after the initial surgery until the end of the study period or death, whichever occurred first. Time to death was calculated as the number of days from the first cataract surgery to death. Participants who did not have a recorded death were censored on April 30, 2019.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew R Rosengart, MD MPH, Principal Investigator — University of Pittsburgh
Locations (1):
- UPMC-Presbyterian Hospital, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after de-identification (text, tables, figures, and appendices) will be shared.
Supporting Information: Analytic Code
Time Frame: Beginning12 months and ending 36 months after publication.
Access Criteria: Data will be shared with researchers who provide a methodologically sound proposal.
  Analyses are limited to those to achieve the aims listed in the approval proposal.
  Proposals should be directed to mrr18@pitt.edu; to gain access, data requestors will need to sign a data access agreement.
  Information regarding accessing data may be obtained after approval of the proposal.